CLINICAL TRIAL: NCT02992171
Title: SHARE - Supportive Care Management for Patients With Hematologic Cancers by Registered Nurses
Brief Title: Primary Palliative Care for Patients With Advanced Hematologic Malignancies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Yael Schenker, MD, MAS, Assistant Professor Director, Palliative Care Research, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PRO16100199; 130225-PEP-16-205-01-PCSM (Other Grant/Funding Number: American Cancer Society)
Record Dates: First submitted 2016-12-07; First posted 2016-12-14 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Advanced Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- care management by oncology nurses (Experimental): The intervention employs a care management approach to facilitate provision of primary palliative care within existing oncology clinic structures. The intervention is deployed through a series of nurse-led encounters occurring before or after regularly-scheduled oncology clinic visits.
  Interventions: Behavioral: care management by oncology nurses

INTERVENTIONS:
Behavioral: care management by oncology nurses — The intervention employs a care management approach to facilitate provision of primary palliative care within existing oncology clinic structures. The intervention is deployed through a series of nurse-led encounters occurring before or after regularly-scheduled oncology clinic visits.

SUMMARY:
This study seeks to develop and pilot-test an oncology nurse-led care management intervention to meet the primary palliative care needs of patients with advanced hematologic malignancies.

DETAILED DESCRIPTION:
Study investigators will develop and pilot-test an oncology nurse-led care management intervention to meet the primary palliative care needs of patients with advanced hematologic malignancies.

Aim 1 is a case series to develop and refine the intervention. During this time, we will develop initial interventionist training materials, study protocols, and a web-based outcomes database; train 2 hematology-oncology nurses; enroll 10 patients with advanced hematologic malignancies and their informal caregivers to receive intervention visits; conduct debriefing interviews; iteratively refine the intervention based on nurse, oncologist, patient, and caregiver feedback; and prepare the protocol for Aim 2. Aim 2 is a pilot study to assess the feasibility and acceptability of administering the intervention and assessing outcomes. We will recruit 30 patients and their informal caregivers to receive the intervention developed in Aim 1 and collect measures of quality of life, symptom burden, anxiety and depressive symptoms, caregiver burden, and healthcare utilization at baseline and monthly for up to three months. Trial outcomes will include: rates of enrollment, study completion, and outcome completion; intervention fidelity; and self-reported measures of study burdensomeness and effectiveness among patients, caregivers, and clinicians.

ELIGIBILITY:
Participants will be (1) patients with advanced hematologic malignancies receiving care at a participating clinic; (2) their caregivers; (3) participating clinicians.

Patient:

Inclusion Criteria:

* adults (≥ 21 years old)
* Refractory or Recurrent hematologic cancer: lymphoma, leukemia, myeloma, amyloidosis (secondary manifestation myeloma & AL Amyloidosis), and CML (CML can only be accelerated or blast phase)
* planning to receive ongoing care from a participating oncologist and willing to be seen at least monthly.

Exclusion criteria:

* chronic myeloid leukemia (CML) OTHER THAN accelerated or blast phase
* unable to read and respond to questions in English
* lacks decision-making capacity, as determined by the patient's oncologist
* unable to complete baseline interview

Caregiver

Inclusion Criteria:

* adults (≥ 21 years old)
* family member or friend of an eligible patient

Exclusion criteria:

* unable to read and respond to questions in English
* unable to complete the baseline interview (patients will be asked to select as caregiver the person who is most likely to accompany them to visits or help with their care should they need it)

Eligible clinicians will be oncology nurses and oncologists practicing at participating clinics.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2020-03-19 (Actual)

PRIMARY OUTCOMES:
Successful enrollment of 30 patient-caregiver pairs | Baseline to 3 months

SECONDARY OUTCOMES:
Consent-to-approach rate | Baseline to 3 months
  Consent to approach rates will be tracked to assess feasibility
Enrolled-to-consent rate | Baseline to 3 months
  Enrolled-to-consent rates will be tracked to assess feasibility
Intervention completion rate | Baseline to 3 months
  Intervention completion rate among enrolled participants will be tracked to assess feasibility
Intervention fidelity | Baseline to 3 months
  Percent of intervention components completed according to protocol will be tracked to assess feasibility
Outcome assessment rate | Baseline to 3 months
  Outcome assessment rates among enrolled participants will be tracked to assess feasibility
Missing data | Baseline to 3 months
  Missing data rates will be tracked to assess feasibility
Acceptability | 3 months
  We will assess acceptability based on patient, caregiver, and clinician responses to closed-end survey questions. Definitions of adequate acceptability based on these surveys include:
  1. > 80% of patient and caregiver participants would recommend the intervention to other patients with advanced hematologic malignancies and their caregivers.
  2. > 80% of patient and caregiver participants agree or strongly agree that intervention visits have been helpful for (a) improving pain or other symptoms, (b) helping with illness understanding, (c) helping with coping, and (d) helping with planning for the future.
  3. > 80% of oncologist participants disagree or strongly disagree that (a) working with intervention nurses has been burdensome or (b) the intervention has been disruptive to clinic workflow.
  4. > 80% of oncologist and nurse participants agree or strongly agree that the intervention (a) has helped me to take better care of my patients and (b) has improved the quality of care.

CONTACTS AND LOCATIONS:
Overall Officials: Yael Schenker, MD, MAS, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share study data with investigators at Duke University. They will have access to de-identified research data, specifically audio recordings and debriefing interviews, for purposes of quality assurance and/or data analysis.

DOCUMENTS (1):
  • Informed Consent Form (2018-09-28): https://cdn.clinicaltrials.gov/large-docs/71/NCT02992171/ICF_000.pdf